CLINICAL TRIAL: NCT00616083
Title: Developing Normative Body Composition Data in Early Infancy
Brief Title: Percent Body Fat in Breast Fed Infants
Acronym: PeaPod
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency); Life Measurement Inc. (Industry); University of Oklahoma (Other); MetroHealth Medical Center (Other); University of Milan (Other)
Responsible Party: Aline Andres, Ph.D / Principal Investiagor, University of Arkansas for Medical Science
Other Study IDs: 56991
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Breast Feeding; Body Composition; Body Fat; Infant; Diet; Healthy Infants
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy breast fed infants

SUMMARY:
The purpose of this study is to learn about normal body composition (% body fat) during the first six months of life in healthy breast-fed babies.

ELIGIBILITY:
Inclusion Criteria:

* Term birth
* Infant must weigh at least 5.5# at birth
* Single birth
* Healthy mother/infant as determined by the investigator
* Intention to breast feed

Exclusion Criteria:

* Significant perinatal morbidity
* Having health, environmental, or economic constraints on growth
* Infants of a mother with diabetes or gestational diabetes

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Helathy breast fed infats, less than a week old living in the Little Rock area.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, Ph.D., Principal Investigator — University of Arkansas
Locations (4):
- United States (3):
  - Arkansas Children's Nutrition Center, Little Rock, Arkansas
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
- Universita degli Studi di Milano, Milan, Italy